CLINICAL TRIAL: NCT01321008
Title: Radiation Therapy Followed by Chemotherapy for Newly Diagnosed Patients With Stage I/II Nasal NK Cell Lymphoma
Brief Title: Stage I/II Nasal NK Cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0035
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2014-05

CONDITIONS: Lymphoma
Keywords: NK cell lymphoma-nasal type; Stage I/II; Radiation therapy; XRT; chemotherapy; CHOP; Cyclophosphamide; Cytoxan; Neosar; Adriamycin; Doxorubicin; Rubex; Vincristine; Oncovin; Prednisone
MeSH Terms: conditions — Lymphoma | interventions — Radiation; Radiotherapy; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation + Chemotherapy (Experimental): Radiation therapy total dose of 50.4 to 54 Gy over 28 to 30 treatments; CHOP Chemotherapy of Cyclophosphamide 750 mg/m2 intravenous piggyback (IVPB), Doxorubicin 50 mg/m2 IVPB, Vincristine 1.4 mg/m2 (max dose 2 mg) IVPB on Day 1, and Oral Prednisone 100 mg daily days 1-5 for four 21-day cycles.
  Interventions: Radiation: Radiation; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Radiation: Radiation — 50.4 to 54 Gy delivered 5 days a week for 28 to 30 treatments.
  Other Names: XRT; Radiation therapy
Drug: Cyclophosphamide — 750 mg/m2 by vein over 1 hour on Day 1 of a 21 day cycle.
  Other Names: Cytoxan; Neosar
Drug: Doxorubicin — 50 mg/m2 by vein over 15 minutes on Day 1 of a 21 day cycle.
  Other Names: Adriamycin; Rubex
Drug: Vincristine — 1.4 mg/m2 (max dose 2 mg) by vein over 15 minutes on Day 1 of a 21 day cycle.
  Other Names: Oncovin
Drug: Prednisone — 100 mg by mouth daily on Days 1-5 of a 21 day cycle.

SUMMARY:
The goal of this clinical research study is to learn if radiation therapy and chemotherapy can help control stage 1 and/or 2 NK cell lymphoma. The safety of radiation and chemotherapy will also be studied.

DETAILED DESCRIPTION:
The Study Treatments:

Radiation therapy is designed to kill cancer cells or to stop cancer cells from growing.

CHOP chemotherapy is made up of the drugs cyclophosphamide, hydroxydaunorubicin (doxorubicin), oncovin (vincristine), and prednisone. It is designed to help control the tumor locally as well as the tumor cells that might have escaped and moved through the body.

Radiation Therapy:

You will receive radiation therapy 5 days a week for 28 to 30 treatments. You will receive a separate consent form that will describe this procedure and its risks in more detail.

Study Visits During Radiation Therapy:

Every week for 6 weeks during radiation therapy:

* You will be asked how you are feeling and about any side effects you may be having.
* Your performance status will be recorded.
* You will have a physical exam.

Chemotherapy Administration:

The amount of time after you finish radiation therapy before you can begin receiving chemotherapy will depend on your recovery time and any side effects you may have. This should be about 3-4 weeks.

On Day 1 you will receive cyclophosphamide by vein over 1 hour, doxorubicin by vein over 15 minutes, and vincristine by vein over 15 minutes. You will take prednisone by mouth on Days 1-5 of each cycle. Each cycle will be 21-days long (or longer if it takes longer for your blood counts to recover). You will receive up to 4 cycles of chemotherapy.

Study Visits During Chemotherapy:

Before Day 1 of Cycle 1:

* You will have a CT scan of head, neck, chest, abdomen and pelvis.
* You will have an Magnetic resonance imaging (MRI) scan of the head and neck.
* You will be asked about any drugs you may be taking and symptoms you may be having.
* Your performance status will be recorded.
* You will have a physical exam, including measurement of your height and weight.
* You will have an echocardiogram (ECHO) and MUltiple Gated Acquisition scan (MUGA) scan.
* You will have an x-ray of the chest.
* You will have an Electrocardiography (ECG).
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If you are able to become pregnant, you will have a blood (about 2 teaspoons) pregnancy test.

On Day 15 of Cycle 1:

* You will be asked about any drugs you may be taking and symptoms you may be having.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 2-4:

* You will be asked about any drugs you may be taking and symptoms you may be having.
* Your performance status will be recorded.
* You will have an ECG.
* Blood (about 2 teaspoons) will be drawn for routine tests.

On Day 15 of Cycles 2-4:

-Blood (about 2 teaspoons) will be drawn for routine tests.

Length of Study:

You may receive radiation and up to 4 cycles of CHOP. You will no longer be able to receive CHOP if the disease gets worse or intolerable side effects occur.

Your participation on the study will be over after the end-of-study and follow-up visits.

Follow-Up and End-of-Study Visits:

If you leave the study early:

* You will have a computed tomography (CT) scan of head, neck, chest, abdomen and pelvis.
* You will have an MRI scan of the head and neck.
* You will have a positron emission tomography (PET)/CT scan.
* Any skin lesions that you may have that are related to the tumor will be measured and photographed.
* You will be asked about any drugs you may be taking and symptoms you may be having.
* Your performance status will be recorded.
* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Routine Follow-up:

* You will also have routine follow-up visits every 3 months for the 1st year, every 4 month during the 2nd year, and every 6 months during the 3rd-5th years. After that, you will have follow up visits 1 time every year. At these visits, the following tests and procedures will be recorded:
* You will have a CT scan of head, neck, chest, abdomen and pelvis.
* You will have an MRI scan of the head and neck.
* You will have a PET/CT scan.
* You will be asked about any symptoms you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Up to 40 patients will take part in this study. All will be enrolled at University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed stage I and II nasal Natural Killer (NK) cell lymphoma.
2. Adequate blood cell counts (i.e. Absolute neutrophil count (ANC)> 1000) at baseline, or willingness to accept supportive measures such as transfusions, filgrastim, and Epoetin. Epoetin will not be administered concurrently with radiation.
3. Patients must have adequate liver function as indicated by: *Bilirubin </= 1.5 times the upper limit of normal (ULN), * Alanine transaminase (ALT) </= 2 times the (ULN) or aspartate transaminase (AST) ≤ 2 times the ULN, *These values must be obtained within two weeks before protocol entry.
4. Patients are required to have adequate renal function as indicated by a serum creatinine </= 2.5 mg/dL.This value must be obtained within two weeks before protocol entry.
5. Left ventricular ejection fraction must be evaluated by nuclear medicine scan or echocardiography and measure >/= 50%.
6. Male patients must agree to use a barrier method of contraception or agree to abstain from heterosexual activity for the duration of the study.
7. Female patients must be willing to use two adequate barrier methods of contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study or be post menopausal (free from menses > two years or surgically sterilized).
8. Female patients of childbearing potential must have a negative serum pregnancy test (BhCG) within 2 weeks of protocol entry.
9. Patients must have the ability to give informed consent.

Exclusion Criteria:

1. Patients with active Hepatitis B and/or Hepatitis C infection.
2. Patients with active infections requiring specific anti-infective therapy are not eligible until all signs of infections are resolved.
3. Patients known to be HIV positive.
4. Patients with pre-existing cardiovascular disease requiring ongoing treatment. This includes: a) Congestive heart failure class III/IV (CHF) per new york heart association (NYHA) criteria. b) Cardiomyopathy, c) Uncontrolled cardiac arrhythmia, d) Unstable angina pectoris, e) Recent Myocardial infarction (MI) (within 6 months).
5. Patients with prior exposure to anthracyclines:
6. Patients who are pregnant or breast-feeding.
7. Patients with psychiatric illness and/or social situations that would limit compliance with the study medication and requirements.
8. Prior radiation to the site of current primary disease, if re-treatment would lead to violation of known radiation dose tolerance limits for that site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina Dabaja, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 20, 2011 to May 8, 2013. All recruitment done at the University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Study was terminated early due to extensive revisions to the study.
Period: Overall Study
Arm/Group | Radiation + Chemotherapy
Started | 1
Completed | 0
Not Completed | 1
Not completed — Early Study Termination | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation + Chemotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) defined as time from treatment initiation day to first documented progressive disease or death due to disease. Reviewed with each 21-day treatment cycle, followed every 3-4 months for first 2 years, annually thereafter.
Time Frame: Day 1 to disease progression or death (up to 5+ years)
Population: Study terminated early, no analysis available.
Arm/Group | Radiation + Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) monitoring during study participation from baseline to completion of 4 cycles, each 21 days. Serious AEs monitored until resolved or clearly determined to be due to stable or chronic condition or intercurrent illness(es).
Description: Collection Period: March 28, 2012 to May 01, 2013.
Arm/Group | Radiation + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation + Chemotherapy (N=1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus Disorder (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination with too small number of subjects to perform analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No